CLINICAL TRIAL: NCT05826912
Title: Multi-Arm Multi-Stage Adaptive Platform Trial (APT) for the Acute Treatment of Traumatic Brain Injury
Acronym: APT-TBI-01
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APT-TBI-01
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Atorvastatin; Minocycline; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention 1: Atorvastatin calcium (ATOR) (Active Comparator): By Mouth (PO) Twice a day (BID) 80 mg/day, with no loading dose, for 28 days
  Interventions: Drug: Atorvastatin Calcium
- Intervention 2: Minocycline hydrochloride (MINO) (Active Comparator): By Mouth (PO) Twice a day (BID) 200 mg loading dose on Day 1, then 100 mg twice daily for 6 days, then placebo twice daily for 21 days
  Interventions: Drug: Minocycline Hydrochloride
- Intervention 3: Candesartan cilexetil (CAND) (Active Comparator): By Mouth (PO) Twice a day (BID) 8 mg once on Day 1, then 16 mg daily for 27 days
  Interventions: Drug: Candesartan Cilexetil
- Matching Placebo (Placebo Comparator): By Mouth (PO) Twice a day (BID) 2 capsules 2x/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin Calcium — Capsule, 80 mg/day, with no loading dose, for 28 days
  Other Names: ATOR
  Arms: Intervention 1: Atorvastatin calcium (ATOR)
Drug: Minocycline Hydrochloride — Capsule, 200 mg loading dose on Day 1, then 100 mg twice daily for 6 days, then placebo twice daily for 21 days
  Other Names: MINO
  Arms: Intervention 2: Minocycline hydrochloride (MINO)
Drug: Candesartan Cilexetil — Capsule, 8 mg once on Day 1, then 16 mg daily for 27 days
  Other Names: CAND
  Arms: Intervention 3: Candesartan cilexetil (CAND)
Drug: Placebo — Capsule, 2x/day for 28 days
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to determine if experimental drug treatment improves recovery after TBI as compared to a control (placebo) group. Changes in recovery will be measured throughout the study. The study drugs listed below are approved by the U.S. Food and Drug Administration (FDA) but are being used "off-label" in this study. This means that the drugs are not currently approved to treat TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-65 years of age, inclusive)
2. Presents to a participating enrollment site and is able to receive first dose within 24 hours of non-penetrating head injury warranting clinical evaluation with a non-contrast head CT based on American College of Emergency Physicians (ACEP) Centers for Disease Control and Prevention (CDC) clinical policy for TBI imaging.
3. Closest, prior to Randomization Glasgow Coma Scale (GCS) score of 9 to 15
4. Acute trauma-related neuroimaging abnormality (subarachnoid hemorrhage, contusion, subdural hematoma, petechial hemorrhage, intraventricular hemorrhage) on cranial CT (CT+)
5. Initial Glial Fibrillary Acidic Protein (GFAP) blood level >100 pg/ml ≤ 15,000 pg/ml determined using a for Research Use Only (RUO) assay(s) or an Investigation Use Only (IUO) assay(s)
6. Persons of childbearing potential (i.e., those not postmenopausal or surgically sterile) may participate provided that they are using adequate birth control methods for the duration of investigational product administration (see manual of procedures for adequate birth control methods)
7. Participants able to undergo Magnetic Resonance Imaging (MRI) scans, no contraindications
8. Participants or legally authorized representative (LAR) willing and able to provide informed consent
9. Participants or LAR able to read, speak, and understand English or Spanish (participating site dependent, where available), including the informed consent form (ICF)
10. Willingness and ability to comply with all study procedures, treatment, and follow-up

Exclusion Criteria:

1. Isolated epidural hematoma
2. Pre-existing conditions including disabling developmental, neurologic, psychiatric, medical disorder that continues to produce functional disability up to the time of injury; or imminent death based on clinical judgement
3. Current enrollment in another interventional study
4. Currently pregnant or currently breastfeeding or planning on becoming pregnant in the next 6 months
5. Current incarceration or in custody
6. Currently prescribed one of the investigational products (or other drugs in the same class) prior to injury; or contra-indicated or as listed in the appendices
7. Hypersensitivity or intolerance to investigational products or the investigational products' respective classes
8. Renal dysfunction (Creatinine Clearance (CrCl) or estimated Glomerular Filtration Rate (eGFR) (<60 mL/minute/1.73 m2)
9. Acute liver disease or hepatic dysfunction (ALT/AST >3 times upper limit of normal lab value)
10. Hemodynamic instability, per participating site physician investigator clinical judgment
11. Inability to swallow investigational product capsule
12. Unable or unwilling to consume animal byproducts, has a gelatin allergy, and/or religious beliefs that do not permit consuming gelatin
13. Intolerance to small amounts of lactose (less than ½ teaspoonful) daily
14. Low likelihood of follow up or study compliance, or any other reason, in the opinion of the participating site investigator, the participants should not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Glasgow Outcome Scale-Extended (GOSE 2-Way) | 2 weeks to 3 months postinjury
  Functional impairment due only to the TBI will be measured using the GOSE Scale-Extended (GOSE 2-Ways). The score ranges from 1-8, with higher scores indicating better recovery. Change will be measured from Week 2 to Month 3 postinjury and compared to placebo.

SECONDARY OUTCOMES:
Change in Blood-based biomarkers (Neurofilament light chain) | Week 2
  Neurofilament light chain (NfL) levels postinjury in participants with TBI will be measured and compared to placebo
Blood-based biomarker (GFAP) | Week 2
  GFAP levels postinjury in participants with TBI as compared to placebo
Imaging biomarkers | 2 weeks to 3 months postinjury
  Comparison of MRI diffusion tensor imaging (DTI) Axial Diffusivity (AD) measure using the average of 4 long association/projections tracts: (i) Anterior Limb of Internal Capsule (ALIC); (ii) External Capsule (EC); (iii) Superior Corona Radiata (SCR); and (iv) Superior Longitudinal Fasciculus (SLF). Change will be measured from 2 Weeks to 3 Months postinjury.
Post-TBI cognitive outcome (BTACT) | Day 3 to Week 4 postinjury
  Neurocognitive impairment due to TBI will be measured using the Brief Test of Adult Cognition by Telephone (BTACT). Change will be measured by composite z-score from Day 3 to Week 4 postinjury
Post-TBI symptom outcome (Rivermead) | Day 3 to Week 4
  Post-concussive symptoms due to TBI as measured by the change in Rivermead Post Concussion Symptoms Questionnaire (RPQ) Total score (0-64) from Day 3 to Week 4. Higher scores indicate more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Manley, MD PhD, Principal Investigator — University of California, San Francisco
Locations (18):
- United States (18):
  - University of California, San Francisco, San Francisco, California
  - Indiana University Health, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Atrium Health Wake Forest Baptist, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas at Austin, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - UTHealth Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - UW Health University Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the Federal Interagency TBI Research (FITBIR) Database.
Time Frame: Shared scientific data will be made accessible as soon as possible, and no later than the time of an associated publication, or the end of performance period, whichever comes first.
Access Criteria: FITBIR qualified investigators will be provided access
URL: https://fitbir.nih.gov/

REFERENCES:
- See also: Related Info — https://tracktbi.ucsf.edu/
- See also: Related Info — https://tracktbi.ucsf.edu/publications
- See also: Related Info — https://tracktbinet.ucsf.edu/